CLINICAL TRIAL: NCT03161145
Title: Treatment Patterns and Outcomes in Unresectable or Metastatic Renal Cell Carcinoma (mRCC) Patients in Japan
Brief Title: A Study to Observe the Treatment Patterns and Outcomes of Patients in Japan With Kidney Cancer That is Unable to be Removed by Surgery or That Has Spread
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-770
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unresectable or metastatic renal cell carcinoma (mRCC): Medical records will be reviewed for treatment patterns and outcomes

SUMMARY:
A medical review chart study in Japan to describe the treatment patterns and outcomes of patients with kidney cancer that is unable to be removed by surgery or that has spread. The clinical data is to be abstracted using electronic data capture (eDC) from patient medical records in Japan.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Adults 20 years and older at the time of initial diagnosis of mRCC
* Alive or deceased as of the date of data collection
* Diagnosis of mRCC between 01-Jan-2012 and 31-Aug-2015

Exclusion Criteria:

* Previously and/or currently enrolled in RCC clinical trials
* Patients have primary cancer other than renal cell cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical records of about 500 patients diagnosed with unresectable or metastatic renal cell carcinoma, including those who have progressed from or discontinued from first-line therapy, between 01-Jan-2012 and 31-Aug-2015 will be enrolled in this study from sites in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Treatment patterns | Approximately 5 years
  measured by retrospective data collection of treatment regimen and duration (including rate of permanent and temporary discontinuation)
Overall survival | Approximately 2 years
  measured by data collection in years
Reason for terminating or switching treatment | Approximately 5 years
  measured by data collection information available in retrospective analysis, if disclosed
Adverse Events | Approximately 5 years
  measured by data collection

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx